CLINICAL TRIAL: NCT04164290
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics of Jiashen Tablets in Healthy Subjects
Brief Title: A Study to Evaluate the Tolerability and Pharmacokinetics of Jiashen Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-JSP-I
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — jiashen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is double-blind with regard to treatment (Jiashen Tablets or placebo) at each dose level. Jiashen Tablets and placebo will be matched for formulation, appearance, and amount. Part B and Part C are open-label with regard to treatment (Jiashen Tablets) at each dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- treatment group 1 (Active Comparator): Jiashen tablet, 0.47g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- treatment group 2 (Active Comparator): Jiashen tablet, 0.94g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- treatment group 3 (Active Comparator): Jiashen tablet,1.88g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- treatment group 4 (Active Comparator): Jiashen tablet,2.82g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- treatment group 5 (Active Comparator): Jiashen tablet,3.76g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- treatment group 6 (Active Comparator): Jiashen tablet,4.23g, oral, once a day
  Interventions: Drug: Jiashen Tablets
- control group 1 (Placebo Comparator): Jiashen placebo tablet,0.47g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo
- control group 2 (Placebo Comparator): Jiashen placebo tablet,0.94g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo
- control group 3 (Placebo Comparator): Jiashen placebo tablet,1.88g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo
- control group 4 (Placebo Comparator): Jiashen placebo tablet,2.82g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo
- control group 5 (Placebo Comparator): Jiashen placebo tablet,3.76g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo
- control group 6 (Placebo Comparator): Jiashen placebo tablet,4.23g, oral, once a day
  Interventions: Drug: Jiashen Tablets Placebo

INTERVENTIONS:
Drug: Jiashen Tablets — 1 tablet
  Other Names: treatment group 1
  Arms: treatment group 1
Drug: Jiashen Tablets — 2 tablets
  Other Names: treatment group 2
  Arms: treatment group 2
Drug: Jiashen Tablets — 4 tablets
  Other Names: treatment group 3
  Arms: treatment group 3
Drug: Jiashen Tablets — 6 tablets
  Other Names: treatment group 4
  Arms: treatment group 4
Drug: Jiashen Tablets — 8 tablets
  Other Names: treatment group 5
  Arms: treatment group 5
Drug: Jiashen Tablets — 9 tablets
  Other Names: treatment group 6
  Arms: treatment group 6
Drug: Jiashen Tablets Placebo — 1 tablet
  Other Names: control group 1
  Arms: control group 1
Drug: Jiashen Tablets Placebo — 2 tablets
  Other Names: control group 2
  Arms: control group 2
Drug: Jiashen Tablets Placebo — 4 tablets
  Other Names: control group 3
  Arms: control group 3
Drug: Jiashen Tablets Placebo — 6 tablets
  Other Names: control group 4
  Arms: control group 4
Drug: Jiashen Tablets Placebo — 8 tablets
  Other Names: control group 5
  Arms: control group 5
Drug: Jiashen Tablets Placebo — 9 tablets
  Other Names: control group 6
  Arms: control group 6

SUMMARY:
Jiashen Tablets as an oral, compound traditional chinese medicine prepatations, have an effect on improvement of the heart failure. This study will assess the safety, tolerability and pharmacokinetics (PK) of Jiashen Tablets, following oral administration of single and multiple ascending dose of Jiashen Tablets.

DETAILED DESCRIPTION:
This study will include a randomized, double-blind, placebo-controlled, single ascending dose design study (Part A), and an open-label SDAD pre-multiple daily ascending dose (MDAD) study (Part B) and an open-label MDAD study (Part C) study.

The study will be conducted in healthy participants and performed at a single study center. 70 healthy participants are planned to be included in the study.

Part A will include six cohorts, 40 participants. Within each cohort, 2 participants will be randomized to receive placebo and other participants randomized to receive Jiashen Tablets. Each participant will receive Jiashen Tablets at the selected dose level or placebo by oral administration in a fasted state once daily.

Part B will include two cohorts, 6 participants, minimum dose group and maximum dose group respectively depending on the findings. Within each cohort, participant will receive Jiashen Tablets at the selected dose level by oral administration in a fasted state once daily.

Part C will include three cohorts, 24 participants. Within each cohort, participant will receive Jiashen Tablets at the selected dose level by oral administration in a fasted state once daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, half male and half female, aged 18-50 years (including the boundary value), the age difference of the same batch of subjects should not exceed 10 years.
2. Have a body mass index of all subjects between 19 and 24kg /m2 (inclusive) and weight of the male subject should be no less than 50Kg and the weight of the female subject should be no less than 45Kg.
3. Passed the smoke test, alcohol and drug abuse test, general physical examination and laboratory examination, chest film, ultrasound, electrocardiogram and other physical and chemical tests.
4. No history of major diseases, no history of smoking and drinking, negative blood pregnancy test of women of childbearing age and no lactation.
5. Obtain informed consent and volunteer to be tested in accordance with the provisions of the Drug clinical trial quality management standard.

Exclusion Criteria:

1. Have primary diseases of cardiovascular，hepatic or renal disease or any other condition. With history of digestive tract diseases, metabolic diseases, and neurological diseases.
2. QTc extension (male >430ms, female >450ms).
3. History of drug allergy or allergic constitution.
4. Family history of hypokalemia, long QT syndrome or other TdP risk factors.
5. Mentally or physically disabled.
6. Any clinically significant abnormalities in physical examination, biochemical and hematuria routine examination, electrocardiogram, chest film and ultrasound examination,.
7. Any positive result on Screening for serum hepatitis B tests (except surface antibodies), hepatitis C antibody , human immunodeficiency virus (HIV) and treponema pallidum antibody test.
8. Those who had taken a drug known to damage an organ within 3 months, taken any drug within 2 weeks, and participated in other clinical trials within 4 weeks.
9. Bleeding tendency.
10. Women during menstruation, pregnancy and lactation.
11. Abnormal vital signs (systolic pressure <90mmHg or >140mmHg, diastolic pressure <60mmHg or >90mmHg;Heart rate <60bpm or >100bpm).
12. Have smoked more than one cigarette per day or used a considerable amount of nicotine products within the previous 3 months, and could not quit smoking during the experiment. Positive screen for the smoke test.
13. Regular drinkers who drank more than 14 units of alcohol per week (1 unit =360mL beer or 45mL spirits with a 40% alcohol content or 150mL wine) during the 6 months prior to the trial, or who tested positive for alcohol, or who do not abstain during the trial.
14. Excessive daily consumption of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250mL) or caffeine test positive.
15. Have a history of blood transfusion or donation in the last 3 months (blood volume greater than 200mL).
16. Have a history of drug abuse and tested positive for drug abuse (morphine, methamphetamine, ketamine, dimethyldimethamphetamine, THC, cocaine).
17. Have a history of antibiotic use in the last month.
18. Have taken lactobacillus products (including yogurt) in the last week.
19. Judgment by the Investigator that the participant should not participate in the study (such as weak, etc).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants. Serious AEs will be recorded from the time of screening.
Number of participants with abnormal blood pressure (BP) | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants. Blood pressure includes both systolic and diastolic BP.
Number of participants with abnormal pulse | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal temperature | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal respiratory | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal findings in 12-lead safety Electrocardiogram (ECG) | From screening (Day-7) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal findings in 24h Holter | From screening (Day -1) till end of trial period
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal physical examination findings | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. The complete physical examinations will include an assessment of the general appearance, skin, cardiovascular, abdomen, head, and neck, lymph nodes, musculoskeletal and neurological systems.
Number of participants with abnormal laboratory assessments: Hematology - absolute count of Red blood cell (RBC), White blood cell (WBC), Platelets | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal laboratory assessments: Hematology-Hematocrit (HCT) | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal laboratory assessments: Hematology - Hemoglobin (Hb) | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal laboratory assessments: Hematology-percentage of Basophils, Eosinophils, Monocytes, Neutrophils, Lymphocytes | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry- Liver function, Renal function, Electrolyte | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants. Liver function: Alanine aminotransferase, Aspartate aminotransferase,Alkaline phosphatase, Gamma-glutamyltransferase,Total Bilirubin, Direct Bilirubin. Renal function: Creatinine,Urea,β2-microglobulin. Electrolyte: Potassium,Sodium,Chloridion,Calcium.
Number of participants with abnormal laboratory assessments: Urinalysis - Urine leukocyte, urine erythrocyte,specific grvity,Glucose, Protein, urobilinogen,bilirubin, ketone, bacteria | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants
Number of participants with abnormal laboratory assessments: coagulation function -Prothrombin Time, Activated Partial Thromboplastin Time,Thrombin Time,Fibrinogen, International Normalized Ratio | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants
Number of participants with abnormal laboratory assessments: Fecal -Fecal Routine and Occult Blood | From screening (Day -1) till follow-up visit (Up to 1 week)
  To investigate the safety and tolerability of Jiashen Tablets following oral administration of single and multiple ascending doses at steady state in healthy participants

SECONDARY OUTCOMES:
Plasma PK analysis: Area under curve at steady state (AUCss) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Maximum observed plasma concentration (Cmax) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Time to reach peak or maximum observed concentration following drug administration (tmax) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Observed concentration at the end of the dosing interval following drug administration at steady state (Cssmin) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Elimination half-life(t1/2) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Maximum observed plasma concentration at steady state (Cmax,ss), time to reach peak or maximum observed concentration following drug administration at steady state (tmax,ss) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Terminal elimination rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve following drug administration (λz) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.
Plasma PK analysis: Terminal half-life, estimated as (ln2)/λz (t½λz) | Day 1,7/8: Pre-dose and 0.5,1.0,1.5,2.0,3.0,4.0,5.0,6.0,7.0,8.0,9.0,10,12,16,24,36,48 hours post-dose and Day 5-6/6-7: Pre-dose
  To characterize the multiple dose PK of Jiashen Tablets and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Tasly Group, Co. Ltd.
Locations (1):
- The second affiliated hospital of tianjin university of traditional Chinese medicine, Tianjin, Tianjin Municipality, China